Organizations

PI (researcher): Pearl McElfish, PhD

# FAMILY MODEL OF DIABETES SELF-MANAGEMENT EDUCATION IN FATH-BASED ORGANIZATIONS

NCT04256486

V.18; 7/18/2024

Organizations

PI (researcher): Pearl McElfish, PhD

# MELELE KO RAORŌK KŌN EKKATAK EO NAETAN "FAMILY MODEL OF DIABETES SELF-MANAGEMENT EDUCATION (DSME) IN FAITH BASED ORGANIZATIONS":

# KEY INFORMATION FOR FAMILY MODEL OF DIABETES SELF-MANAGEMENT EDUCATION (DSME) IN FAITH BASED ORGANIZATIONS:

Kōmij kajjitōk bwe kwōn kelet elañe kwōj kōnaan ak jab kōnaan bōk konaam ilo ekkatak in ñan jibañ armij ro ewōr aer nañinmej in tōñal koba baamle ko aer ñan katak kōn nañinmej in tōñal im wāwein ko ñan kōjparok. Kilaaj ko an ekkatak in renaj kōmman ilo imōn jar ko ak jikin ko jet an mwōn jar ko.

Pepa in ej kwalok melele ko raurōk ñan jibañ iok kōmman kelet eo am im kalikar kwōj ke bōk konaam. Emōj droor melele ko remelijlok ālikin pepa in. Lelok kajjitōk ko am ñan team eo ej bōk eddoin ekkatak in. Elañe ewōr am kajjitōk tok ālik, melele ko ñan tōbar rijerbal ro an ekkatak in rej bed āliktata in pepa kein.

We are asking you to choose whether or not to volunteer for a research study about helping persons with diabetes and their family members learn how to manage diabetes. Classes for this study will be done in a church or other faith-based setting.

This page gives you key information to help you decide whether to participate. We have included detailed information after this page. Ask the research team questions. If you have questions later, the contact information for the research investigator in charge of the study is below.

# EKKATAK IN EJ KŌN TA IM EWI AITOKAN? WHAT IS THE STUDY ABOUT AND HOW LONG WILL IT LAST?

Ilo ad kōmmane ekkatak in, jej kōjatdikdik ke jenej maroñ loe elañe Rimajōl ro ewōr aer nañinmej in tōñal remaroñ kōkmanman lok ejmour ko aer im jokkin mour ko aer elañe er im baamle ko aer renej ekkatak ibben dron kōn bōbrae nañinmej in tōñal ko aer. Jej bar kōnan jelā elañe katakin kōn nañinmej in tōñal ilo mwōn jar ko emman lok jen jikin ko jet. Nān kajjioñ men in, jenej etale elañe nañinmej in tōñal ko aer rej emman lok. Ewōr 408 rutto in Majōl ro (18 iiō im rutto lok) im ewōr aer nañinmej in tōñal im 1-2 uwaan baamle ko aer renej maroñ mōttan ekkatak in. Ilo am bōk konaam ilo ekkatak in eo aitokan enej tarrin 10 allōñ ñan juōn iiō koba 10 awa in ekkatak kōn nañinmej in tōñal ilo 8-12-wiik aitokan im konej bar bōk konaam ilo jillu nān emen ien ko nān ebbōk melele ko am. Nē konej kobatok ilo ekkatak in, renej kajjitōk ibbam nān bed ilo kilaaj in kejbarok nañinmej in tōnāl ko im ien ebbōk melele ko ijo renej ebbōk melele ikkijen ejmour jen kwe.

By doing this study, we hope to see whether Marshallese patients with diabetes can improve their health and quality of life if they and their families learn together about managing their diabetes. We also want to learn if teaching about diabetes in a church setting is better than teaching in other places. To test this, we will measure if their diabetes improves. Up to 408 Marshallese adults (ages 18 years and older) with diabetes and one to two of their family members may be part of this study. Your participation in this research will last about 10 months to one year with 10 hours of diabetes education over an 8-12 week period and you will participate in three to four

Organizations

PI (researcher): Pearl McElfish, PhD

data collection events. If you join the study, you will be asked to attend diabetes management classes and data collection events where we collect health information from you.

# ETKE INEJ MAROÑ KELET BWE IN BŌK KONAŌ ILO EKKATAK IN? WHY MIGHT I CHOOSE TO VOLUNTEER FOR THIS STUDY?

Emōj kajjitōk ibbam nan koba tok ilo ekkatak in konke ewor am naninmej in tonal ak konke juon eo uwaan baamle eo am ewor an naninmej in tonal ej kur tok eok nan koba tok ibbeir. Einwot juon eo ej bed ilo ekkatak in, konej bed ilo kilaaj in tonal kein ko rej komman jen juon eo ewor an kapeel ikkijen katakin kon naninmej in tonal. Ilo ien kilaaj kein kwonej ekkatak kon kejbarok ad mona, makutkut, etale tonal eo am, im kapeel ko jet im rej jiban armej bobrae naninmej in tonal. Am bed ilo ekkatak in emaron jiban bwe kwon ejmour lok, im emaron jiban armij ro ewor aer naninmij in tonal iliju im jeklaj. Nan melele ko remelijlok ikijien emman ko an ekkatak in, kwonaj riiti pepa in Full Consent eo elikin pepa in.

You are being invited to join in this study because you either have diabetes or because a family member with diabetes has invited you to join with them. As a person in the study, you will attend diabetes education classes led by a trained diabetes teacher. During these classes you will learn about healthy eating, being active, tracking blood sugar, and other skills that help people to manage diabetes. Being in the study may help your health improve and may help other persons with diabetes in the future. For a complete description of benefits, refer to the Full Consent.

# ETKE INEJ KELET BWE IN JAB BŌK KONAŌ ILO EKKATAK IN? WHY MIGHT I CHOOSE NOT TO VOLUNTEER FOR THIS STUDY?

Emaron wor ien eo im juon armij emaron jela kon melele ko ikijen ejmour eo am, botaap jenaj kojparok bwe en jab walok wawein in. Ilo am bok kilaaj ko, armij ro jet remaron jela melele ko kon kwe make elane kwonaj kenono kaki.

Ejjelok kallimur ke ekkatak in enaj jibañ eok. Nan melele ko remelijlok ikijien emman ko an ekkatak in, kwonaj riiti tarlepen pepa in Mālim eo ālikin pepa in.

There is the chance that someone could find out about your private health information, but we will take special care to reduce this risk. By taking part in the educational sessions other people in the session may learn information about you if you talk about yourself.

There is no guarantee that the study will help you. For a complete description of risks, refer to the full Consent.

Organizations

PI (researcher): Pearl McElfish, PhD

# IJ KE AIKUJ BŌK KONAŌ ILO EKKATAK IN?

### DO I HAVE TO TAKE PART IN THE STUDY?

Jaab. Ejjelok bwōd ne kwonaj ba jaab. Elane kwonaj errā in bōk konaam ilo ekkatak in, ej aikuj kōnke kwe make kwōj kōnaan bōk konaam. Eban jako jabdrewōt maron ko am ak jiban ko ekkā am būki elane kwonaj kelet in jab bōk konaam.No. It is okay to say no. If you decide to take part in the study, it should be because you really want to volunteer. You will not lose any services, benefits, or rights you would normally have if you choose not to volunteer.

Organizations

PI (researcher): Pearl McElfish, PhD

# **University of Arkansas for Medical Sciences Informed Consent Form**

Jej kajitōk ibbam bwe kwōn bed ilo ekkatak in. kwojjab aikuj bed elañe kwojjab kōnan. We are asking you to be in a research study. You do not have to join the study.

o Kwōj maron wōt bōk jiban ikkijen taktō jen UAMS mene kwojjab bed ilo ekkatak in. You can still get your medical care from UAMS even if you are not in the study.

Jouj im bōk ien elap joāan wōt eo kwoj aikuji āan riiti pepa in im kelet ta eo emman nan kwe. Please take as much time as you need to read this form and decide what is right for you.

# Etke rej kajjitōk ibba bwe in bed ilo ekkatak in?

Why am I being asked to be in this research study?

- Jej konan katak elap lok kon katakin kojebarok naninmej in tonal. We want to learn more about teaching diabetes self-management.
- Ekkatak in enej jiban koj jela elaplok melele ko elane rimajol ro ewor aer naninmej in tōnal im remaron kōkmanmanlok ejmour ko aer im wāwein jokkunmour ko aer elane er im baamle ko aer renej ekkatak wāwein kojebarok naninmej in tonal ko aer ilo mwon jar ko. This study will help us learn more about whether Marshallese patients with diabetes can improve their health and quality of life if they and their family learn about managing their diabetes in a church setting.
- Kōmij kajjitōk ibben armej einwōt kwe eo im ewōr an naninmej in tōnal ak emōj kūr tok eok jen juon ian baamle eo am ewōr an nañinmej in tōnal nan jiban kōm. Ewōr 408 rutto in Majōl ro (18 iiō im rutto lok) im ewōr aer naninmej in tōnal im juon ian baamle ko aer bwe ren bar mottan ekkatak in. We are asking people like you who have diabetes or have been invited by a family member with diabetes to help us. Up to 408 Marshallese adults (ages 18 years and older) with diabetes and one of their family members may be part of this study.

Version #: 18 IRB# 229034 Date: 20240718 Page 5

Organizations

PI (researcher): Pearl McElfish, PhD

# Elane ewor jabdrewot men eo ijjab melele kake?

# What if I don't understand something?

- Emaron wor melele ko kwojjab melele kaki ilo pepa in. Elane kwoj konaan, ro rej jerbal ilo ekkatak in remaron riiti im etale pepa in ibbam. This form may have words you don't understand. If you'd like, research staff will read it with you.
- Kwomaron komman am kajitok jabdrewot ien mokta, ien eo, ak ālikin ekkatak in. You are free to ask questions at any time before, during, or after you are in the study.
- Jouj im kajjitōk joñan wōt eo kwoj kōnan mokta jen am kelet elañe kwoj kōnan bed ilo ekkatak in. Please ask as many questions as you like before you decide whether you want to be in this study.

# Ta enej walok elañe inaj ba aet, ij kōnan bed ilo ekkatak in? What will happen if I say yes, I want to be in this study?

Jenaaj lale mokta elane kwoj ekkar nan bed ilo ekkatak in. Jenaj kajjitok ibbam elane kwe...We first will see if you qualify to be in the study. We will ask if you...

- juōn ri Majōl, identify as Marshallese.
- 18 am iiō ak rutto lok, are 18 years or older.
- ewōr nañinmij in tōñal type 2 ibbam ak juon eo uwaan baamle eo am ewōr an nañinmej in tōñal type 2 (HbA1c eo ej einwōt ak laplok jen 6.5), have type 2 diabetes (HbA1c equal or greater than 6.5) or are a family member of a person with type 2 diabetes.
- emōj am bōk kilaaj in DSME ilowaan iiō ko lalem rej mootlok, have received DSME in the past five years.
- ewōr juōn armij uwaan baamle eo am im emōj an errā in bōk konaan ilo ekkatak in ibbam, have at least one family member who will agree to take part in the study with you.
- Kwōj lōmnak in emmakit jen jikin ko rej kōmmane ekkatak eo ie ilowaan 12 allōn̄ ko, Plan to move out of the area in the next 12 months
- Ewor am nañinmej ko renej bobraik eok jen am bed ilo kilaaj ko einwot nañinmej ko ejjelok unokaer ak rejjab maroñ komadmodi, jab maroñ jutak make ian ak ejjab maroñ etetal, nañinmej in komalij, jab lolok ijen ak jaroñroñ, ak ejjab jejjet wawein aer moña, have an illness that would prevent you from fully participating in the classes such as terminal illness, non-ambulatory, severe mental illness, severely impaired vision or hearing, or eating disorder

Elañe kwoj ekkar nan bōk konaam, kōm naj kōmmani wāwein kein:

If you qualify, we will do these things:

Organizations

PI (researcher): Pearl McElfish. PhD

> Kadeloñ etam ilo kilaaj in nañinmij in tōñal ko. Kilaaj ko ikijien nañinmej in toñal renaaj 10 awa aitokier ilowaan 8-12 wiik. Im kajojo ijen kilaaj kein enaj 60 nan 90 minit aitokier. Kilaaj ko renaj kōmman ilo mwōn jar ko ak bar juōn jikin an mwōn jar ko. Ro rej bōk konaer im uwaan baamle ko aer renej bed ilo kilaaj kein ilo juon doulul in armej ibben ro jet mõttan ekkatak in im ro uwaan baamle ko aer. Ne kwoj konaan tobar eok ilo text message ak jeje waj ilo cellphone eo am, jenej jeje waj ilo kajojo wiik nan kakemejmej eok kon ien eo, awa eo, im ia eo kilaaj eo enej komman. Jeje waj ak text message ekoba juon link eo enej boklok eok ñan calender eo ej kallikar kilaaj ko an mwon jar eo am. Jenej maron bar jeje waj nan kakemejmej eok kon raan in data collection ak ebbōk melele ko. Nan ad maron nej jeje wōj nan cellphone ne am, jenej lelok nōmba in cellphone eo am n̄an Twilio. Ejjelok bar jabdrewōt melele jenej lelok n̄an Twilio. Ilo kilaaj kein, kwonaj ekkatak kon wawein kojebarok am mona, makutkut im exercise, etale joñan tōñal, im wāwein ko jet remaron jiban ikijien naninmej in tōñal. Jenaj bar kajjitōk ibben armij ro nukum kwar kūr er bwe ren bar bōk konaer ilo kilaaj ko ikijien nañinmij in tōnal. Armij ro nukum remaron bed ilo kilaaj ko, jekdron ne raar jab lelok etaer nan ekkatak in. Enroll you in diabetes education classes. Classes will cover 10 hours of diabetes education over an 8-12 week period and each class will last between 60 and 90 minutes. Classes for this study will be done in a church or other faith-based setting. Participants and family members will attend classes in a group setting with other participants and their family members. If you agree to be contacted via text message, we will text you each week during classes to remind you of the date, time, and location of your class. Class reminder texts may include a link leading to a class calendar for your church. We may also text you to remind you of upcoming data collection events. In order to contact you via text message, we will share your phone number with the third-party service Twilio. No other information will be shared with Twilio. During these classes you will learn about healthy eating, being active, tracking blood sugar, and other skills that help people to manage diabetes. The family members you invite will be asked to join the study and participate in diabetes education classes. Family members can attend the classes, even if they are not in the study.

- Jenaaj kajjitōk kōn melele ko am einwōt etam, atōreej in jikin jokwe, talepon nōmba, raan in lotak, kōrā/emmaan, mare, kabijuknen, jikuul, jerbal, injuren, taktō, im jikin ko kwōj itok jeni. Jenaj kajitōk kōn melele ko ikijien ejmour, einwōt jonan aitok, eddo, bōroro, kakōlkōl in tōnal, aibōlat, jiban jen baamle eo am, exercise ak makūtkūt, kain uno ko kwōj būki, mōnā, dren, im melele ko ikijien am kiki. Ask about demographic information such as your name, address, phone number, date of birth, sex, marital status, number of persons in your home, education, employment, insurance status, ability to access health care, and race/ethnicity. Ask about information related to your health such as height, weight, pregnancy status, tests for diabetes, blood pressure, support from your family, managing your weight, exercise, what medications you take, what you eat and drink, and your sleep.
- Rijerbal ro rej kajin majol renaj riiti kajjitok ko im kanne pepa in ibbam, ne kwoj konaan. Kwōjjab aikuj uwaak jabdewōt kajjitōk elañe kwojjab kōnaan. Bilingual staff members will read the questions out loud and fill out the form with you, if you like. You don't have to answer any questions you don't want to answer.

Version #: 18 IRB# 229034 Page 7

Organizations

PI (researcher): Pearl McElfish, PhD

Kajojo mwōn jar ko renaj maroñ bed ilo juon ian doulul ko ruo. Mwōn jar ko ilo doulul eo juōn renaj mōkaj im jino kilaaj ko aer ālikin wōt aer ebbōk melele ko aer. Mwōn jar ko ilo doulul eo kein karuo renej bōk ejja kilaaj ko wōt bōtaab renaj jino ālikin doulul eo juōn.

Jenaj ebbōk melele (data collection) jen kwe im ro nukum raar errā in bōk konaer ilo ien kein: mokta jen an jino kilaaj kein, ālikin an jemlok kilaaj eo eliktata, im 3 allōn ālikin kilaaj kein. Melele ko jenaj aini ilo ien data collection ko renaj einwōt kein: jonan aitokam, eddoūm, im blood pressure ak aibōlat. Kwe im ro nukum rej bed ilo ekkatak in naj bar lale jonan tōnal ko aer. Kakōlkōl kein renaj aikuj bwe jen wākār jabon adiin peim im bōk jidrik bōtōktōk. Ilo ruo lak nān jilu iaan iien data collection kein, kwe im eo uwaan baamle eo am naaj bareinwōt kanne survey ko rej kajjitōk kōn naninmij in tōnal im wāwein kōjbaroke. Ilo kajojo ien data collection kein 3 ak 4, renaj bōk tarrin 2-4 awa aitokier.

Each church will be assigned to one of two groups. Churches in one group will begin classes immediately after the first data collection event. Churches in the second group will have the same classes but they will start later than the classes for the first group.

Before classes begin, after classes end, and 3 months after the classes, we will collect information from you and your participating family members. These data collection events will include measuring your height, weight, and blood pressure. You and any participating family members will also have some tests done to track blood sugar over time. This test will require a finger prick to get a small drop of blood. At two to three of the data collection events, you and any participating family members will also fill out surveys that ask questions about diabetes care and management. Each of the 3-4 data collection events will last about 2-4 hours.

# Ewi aitokan ekkatak in?

How long will this study take?

Elañe kwonaj errā nan bed ilo ekkatak in, konaj bok tarrin 10 awa in kilaaj in tōnal, 8-12 wiik aitokan im bōk konaam ilo 3-4 ien ebbōk melele ko ak data collection. Aolepen ekkatak in, koba kilaaj in tōnal ko im ien data collection ko, emaron bōk jonan in 10 allōn nan juon iiō aitokan.

If you agree to join this study you will participate in 10 hours of diabetes education over an 8-12 week period and you will participate in three to four data collection events. The entire study including, the diabetes education classes and data collection will be over a period of about 10 months to one year time period.

# Ak ne inaj ba jaab, ijjab konaan bed ilo ekkatak in?

What if I say no, I do not want to be in this study?

Ejjelok jorāān enaj walok. Nothing bad will happen.

Family Model of Diabetes Self-Management Education in Faith Based Organizations Pearl McElfish, PhD Study Title:

PI (researcher):

Kwonej maron wot bok jiban ikkijen takto ilo UAMS. You can still get medical care at UAMS.

Version #: 18 IRB# 229034 Date:20240718 Page 9

Organizations

PI (researcher): Pearl McElfish, PhD

### Ewor ta elane inaaj ba aet, im ukot ao lomnak tok alik?

# What happens if I say yes, but change my mind later?

- Komaron bojrak jen ekkatak in jabdewot ien. You can stop being in the study at any time.
- Ejjelok jorāān enaj walok. Nothing bad will happen.
- Kwōj maron wot takto ilo UAMS. You can still get medical care at UAMS.
- Elañe kwōj lōmnak in bōjrak jen ekkatak in, call e Dr. Pearl McElfish ilo 479-713-8680 If you decide to stop being in the study, call Dr. Pearl McElfish at 479-713-8680.

#### Ewor ke onāān ao bed ilo ekkatak in?

# Will it cost me anything to be in the study?

Ejjelok onāān am bed ilo ekkatak in.

The study will not cost you anything.

# Enaaj ke wor ao kolla kon ao bok konao ilo ekkatak in?

# Will I be paid for being in the study?

Aet. Kōm naj lewaj \$20 – \$100 gift card nan kamolol eok kōn ien ko am. Ilo jilu nan emen ien ebbōk melele kein jenaj jone aitokam, eddoum, aibōlat, im bōk jidik bōtōktōk nan lale jonan tōnal eo am iumwin 3 allōn ko. Ruo lak nan jilu iaan iien data collection kein enaj bareinwōt wōr juon survey, nan iien kein kom naaj lewaj nan eok \$30 gift card nan pre-intervention im \$100 ilo gift card ilo ien ebbok melele kein 2 alikin kilaaj im mokta jen an jinoe kilaaj ko nan ro rej bed ilo kilaaj ko emokaj aer jinoe im ro rej bed ilo kilaaj ko erumwij aer jinoe. Kwoban bōk onāām jen am bed ilo kilaaj ko. Elañe kwonaaj bed ilo aolepen jilu ñan emen ien ebbōk melele kein (data collection), kwonaj bōk jonan in \$150 nan \$180 ilo gift card. Konej maron in wot ebbōk gift card ilo am nej bed ilo ien data collection ak ebbōk melele ko. Armej ro renej bed ilo 6 iaan ien ekkatak ak kilaaj ko 8 naaj bar lelok nan er \$100 gift card. Ne kwonaaj ped ilo jilu nan eman ien data collection ak ebbōk melele ko im 6 ian kilaaj ko, kwonaaj maron bōk jonan in \$250 nan \$280 ilo gift card. Nan am bok kollā kein, jenej kajjitok ibbam bwe kwon kadede lok pepa in gift card eo koba lok survey eo nan kallikar etam im signature eo am. Melele kein renej kakuni ilo juon jikin eo etiljek ilo UAMS im rijerbal ro wot ilo ekkatak in nej maron delone. Et eo etam jenij tilmake lok nan Tango Rewards Genius eo, ro rej loloodjake kaat in jiban ko. Ejjelok bar melele ko ikkijem ilo pepa in ijellokin wot etam ak jabdrewot uwaak in melele ko am ilo ekkatak ko jar jerbal ibbam kaki jenej lelok nan Tango Rewards Genius eo.

Yes. We will give you a \$20-\$100 in gift cards to thank you for your time. At three to four data collection events we will collect your height, weight, blood pressure, and prick your finger to collect HbA1c. For those shorter data collection events, we will give you \$20 in gift cards. Two

Organizations

PI (researcher): Pearl McElfish, PhD

to three of the data collection events will also include a survey, for those data collection events we will give you \$30 in gift card for pre-intervention and \$100 gift card for data collection events immediate post and pre intervention #2 for those who are in the intervention arm and waitlist arm respectively. You will not be paid to attend the educational classes. If you attend all three to four information collection events, you will receive \$150 to \$180 in gift cards. You will only receive gift cards for the times you attend the events. Persons who attend at least 6 of the 8 educational sessions will receive an additional \$100 gift card. If you attend all three to four data collection events and at least 6 of the classes, you will receive a total of \$250 to \$280 in gift cards. To receive payment, we ask that you complete a Gift Card Receipt Form following the survey which records your name and signature. This information will be kept on a secure UAMS server and only the program staff will have access to the information. Your name will be shared with Tango Rewards Genius, the gift card vendor. No other information from the gift card form will be shared with Tango Rewards Genius.

# Ekkatak in enaj ke jiban na ilo jabdewot wawein?

#### Will being in this study help me in any way?

Ekkatak in emaron ak emaron jab jiban eok, botaab emaron jiban armij kojbarok naninmij in tonal Type 2 ilju im joklaj.

Being in the study may or may not help you but may help people manage their Type 2 Diabetes in the future.

#### Ta kauwōtata ko remaron walok jen aō bed ilo ekkatak in?

What are the risks of being in this study?

#### Kauwotata ko rej:

The risks are:

- Kauwotata ko ekkā aer walok jen raan nan raan. The risks for this study are no more than what happens in everyday life.
- Komaron abonono ilo aer wākāre addin bweum. You may experience discomfort from the finger prick.
- Ro jet remaron jelā ke kwoj bed ilo ekkatak in im jelā melele ko am im kwojjab konan bwe ro jet ren jelā. Kom nej kajjion jonan wot am maron kojebarok melele ko am, einwot an komeleleik elap lok ijiko tok imaan ilo pepa in. Someone could find out that you were in the study and learn something about you that you did not want others to know. We will do our best to protect your privacy, as explained in more detail later in this form.
- Ilo am naj bed ilo kilaaj ko, armij ro jet ilo kilaaj eo remaroñ roñ melele ko am elañe konaaj kenono kōn kwe make. By taking part in the educational sessions other people in the session may learn information about you if you talk about yourself.

Organizations

PI (researcher): Pearl McElfish, PhD

# Elane inaaj naninmej ak joraan ilo ao bed ilo ekkatak in?

# What if I get sick or hurt while I'm in this study?

Elañe kwonaaj jorāān ilo ien eo kwoj bed ilo ekkatak in, jenaj jibañ eok kabbok jibañ eo kwoj aikuji. Ekoba first aid, jikin taktō ko rediñ, im jikin takto ko jet. If you get hurt when you are here for the study, we will help you get the care you need. This may include first aid, emergency care, and/or follow-up care.

# Ta wāwein ko jet ijjelokin bed ilo ekkatak in?

# What are the alternatives to being in this study?

Kwomaron jab bed ilo ekkatak in.

Ejjelok bar jet wāwein ko jet nan bed ilo ekkatak in, einwot an jab komman komadmod ak wāwein ko jet remaron jiban eok.

You do not have to be in this study.

There are no alternatives to being in this study, as it does not involve treatment or other procedures that may help you.

# Remaron ke jolok na jen ekkatak in elane ij konan wonmaanlok wot?

### Can I be taken out of the study even if I want to continue?

Aet, taktō eo (ak eo ej bōk eddoin ekkatak in) remaroñ kabōjrak am bōk konaam ilo ekkatak in elañe:

Yes, the study doctor (or head researcher) can take you out of the study if:

- Kwojjab loori kõmelele ko an ekkatak in. You do not follow study instructions.
- Ejjab ekkar im emman ñan kwe bwe kwōn wōnmaanlok wōt. It is not in your best interest to continue.
- Ekkatak in enaaj bojrak kon jabdrewot wun. The study is stopped for any reason.

### Melele ta ko renaj būki jen na ilo ekkatak in?

### What information will be collected about me in the study?

Ilo ekkatak in, jenaj aikuj melele ko kōn kwe, einwōt:

During the study, we will need to learn private things about you, including

 Melele ko am einwöt etam, atöreej, talpoon nömba, im melele ko jet rej kallikar wön kwe. General contact and background information about you, such name, address, telephone number, and other demographic information

Organizations

PI (researcher): Pearl McElfish, PhD

Melele ko ikijien ejmour, einwöt joñan aitok, eddo, böroro, kakölköl in töñal, aibölat, jibañ jen baamle eo am, makütküt ak exercise, wuno ta ko kwöj büki, im möñā ko kwoj kañi koba dren ko nimöm. Medical information about you, such as height, weight, pregnancy status, tests for diabetes, blood pressure, support from your family, managing your weight, exercise, what medications you take, and what you eat and drink

Ne kwoj rinañinmej ilo jikin taktō eo an UAMS, jenej kajjitōk mālim eo am ñan ad maroñ bōk melele ko am kōn tōñal jen jikin taktō eo am ilo nej tarrin 12 allōñ ālikin kilaaj ko, ilo nej 18 allōñ ālikin kilaaj ko, im ilo 24 allōñ ālikin kilaaj ko. If you are a patient of UAMS, we will request permission to get information about your diabetes care from your healthcare provider 12 months after classes, at 18 months after the end of the classes, and at 24 months after the end of the classes.

# Won enaj loi melele kein? Ewi wawein am nej kojbaroki jen ro jet?

# Who will see this information? How will you keep it private?

- Team eo loloodjake ekkatak in enej jelã etam im naaj loi melele ko am. The local study team will know your name and have access to your information.
- Enej et eo etam wot jenej tilmake lok nan Tango Rewards Genius eo, ro rej lolodjake kaat in jiban ko. Only your name will be shared with Tango Rewards Genius, the gift card vendor.
- Jenaj loloodjake im kojbarok bwe ro rejjab bed ilo ekkatak in ren jab loi melele ko am. We will do our best to make sure no one outside the study knows you are part of the study.
- Jeban likit etam ilo melele ko am jenej buki jen kwe ilo ien ekkatak in. We will take your name off of information that we collect from you during the study.
- Ne jenaj kwalok tōbrak ko an ekkatak in ilo pepa ko an university ko, jeban likit etam ak jabdrewōt melele ko renaj kallikar wōn kwe. When we share the results of the study in academic publications, we will not include your name or anything else that identifies you.
- Ewōr armij ro rej loloodjake bwe en jimwe an ettōr ekkatak in. Armij rein remaron loi melele ko am. Armij rein rej There are people who make sure the study is run the right way. These people may see information from the study about you. They are
  - ✓ Rijerbal ro an ekkatak in, The research staff
  - ✓ OHRP (Office for Human Research Protections), juon federal agency, OHRP (Office for Human Research Protections), a federal agency
    - ✓ UAMS Institutional Review Board, UAMS Institutional Review Board
    - ✓ Obiij ko rellaplok im rej etali jerbal kein, Other institutional oversight offices

Kakien ko an State aikuj bwe jen ba ñan ijoko rej eddoik elañe jejlā, State law requires we tell the authorities if we learn

Organizations

PI (researcher): Pearl McElfish, PhD

✓ Kōn kakure ko nan ajiri ak rutto ro, about possible child or adult abuse

✓ Elane komaron kakure eok make ak ro jet, that you might hurt yourself or someone else

# Melele ko aō renaj bed ia im ewi toon aer naj dābiji?

# Where and how long will my information be kept?

- Jenaj droor jet nomba ko renaj bok jikin etam im droor melele ko am ilo juon jikin kakkon eo etiljok. We will code your information and keep the key to the code in a locked file on a secure UAMS server.
- Rijerbal ro wot rekkar ilo ekkatak in remaron jela nomba ta ko rej kallikar melele ko am. Only designated research study staff will be able to link your information to you.
- Ilo nej dedelok in ekkatak in, melele ko am naj jako im nomba ko nan melele ko am renej juloki. At the conclusion of the study, the data will be permanently de-identified and the key code will be destroyed.
- Melele ko am renaj jako ālikin jiljilimjuon iiō ko ālikin an jemlok ekkatak in elañe kwonaj kwalok am jab kōnaan bwe jen kōjerbal melele ko am ñan ekkatak ko jet ilju im jeklaj. Your de-identified information will be destroyed seven years after the end of the research if you don't agree to let us keep your information for future research.

Elañe inaaj bōjrak jen ekkatak in, ta enaj walok ñan melele ko aō im emōj kar būki ilo ekkatak in?

If I stop being in the study, what will happen to any information collected from me in the study?

Jenaaj komakit melele ko am jen ekkatak in elane kwonaj ba jen jab kojerbali. Jejjab maron komakit melele ko am jen ekkatak in alikin an moj ad jeje pepa ikijien ekkatak in. We will remove your data from the study if you tell us you want it removed. We will not be able to take your information out of the study after it has been published.

Melele ko aō ak teej ko aō jen ekkatak in renaj ke kōjerbali nan jabdrewōt wāwein ko jet, koba nan ekkatak ko ilju im jōklaj?

Will my information or samples from the study be used for anything else, including future research?

• Aet. Elañe kwonej errā ijin ilal, jenej kōjerbal melele ko am ñan ekkatak ko ilju im jōklaj ikijien nañinmij in tōñal im nañinmij ko jet aeirlok wōt. Yes. If you agree below, we will use the information in future research related to diabetes and other metabolic disease.

Organizations

PI (researcher): Pearl McElfish, PhD

Melele ko kōn kwe renaj kōmakiti im juon code ak nōmba ilo juon key nan code eo nan kōjenokloki. Melele ko renej kakuni ilo juon file eo ej lock im etiljok ilo UAMS ekkar nan kakien ko an UAMS. Melele ko ilo computer ewor aer password im ejjab aolep rijerbal ro an ekkatak in remaron deloni. Elane kwonaj ukot am lomnak kon kojerbal melele kein am nan ekkatak ko iliju im joklaj, kūr lok Dr. Pearl McElfish ilo 479-713-8690 ak ilo pamcelfish@uams.edu. Personal identifiers will be removed and a special code or number with a key to the code will be kept separately. Information will be stored in a locked file on a secure UAMS server consistent with UAMS policies. Electronic data will be in a password protected database with access restricted to research staff. If you change your mind about use of your information in future studies, contact Dr. Pearl McElfish at 479-713-8690.

- Jeban aji melele ko am ñan armij ro jet ijjelokin rijerbal ro ilo ekkatak in. Your information will not be shared with persons other than the current research staff.
- Elañe kwonaj errā bwe jen kōjerbal melele ko am ñan ekkatak ko ilju im jeklaj, innem melele ko am renaj bed wōt iumwin kōjparok ko an UAMS. If you agree to let us keep your information for future research, we will keep it indefinitely.
- Elañe kwojjab errā bwe jen dābij melele ko am ñan ekkatak ko ilju im jeklaj, innem jenaj julok aolep melele ko am jiljimijuon iiō ālikin an jemlok ekkatak in. If you don't agree to let us keep your information for future research, your information will be destroyed seven years after the end of the research.

# Kom nej ke ba nan na kon tobrakin ekkatak in?

Will you tell me the results of the study?

• Aet. Jenaaj kennanik eok im kajojo armij ro rej bed ilo ekkatak in kon jabdrewot melele ko reaurok renaj walok jen ekkatak in. Yes. We will tell you and every person in the study about anything important that we discover from the study.

Kom nej ke konnanok iio kon jabdewot wawein ko remaron jelet ejmour eo ao?

Will you tell me anything you learn that may impact my health?

Aet. Jenaaj k\u00f3nnan\u00f3k eok ela\u00eae enaaj walok jabdew\u00f3t melele ko raur\u00f3k ikijien ejmour eo am. Yes. If we learn something about you that might be important for your health, we will tell you.

Ta enaaj walok elane ewor melele ko rokaal ikijien ekkatak in?

What if new information comes up about the study?

Organizations

PI (researcher): Pearl McElfish, PhD

Jöknaan bwe kwon jelä kön jabdewöt melele ko im remaron jäniji am lömnak kön am bed ilo ekkatak in. We want you to know about anything that may change your mind about being in the study.

- Team eo ej loloodjake ekkatak in enaaj konnanik eok ilo an: The study team will let you know by:
  - ✓ call eok, calling you
  - ✓ jilkinwaj juon leta, sending you a letter
  - ✓ kōnnanik eok ilo juon ian ien bar rool waj ko, telling you at a follow up visit

# Ak ne ewor ao kajjitok?

# What if I have questions?

- Kūr lok armij eo ej bõk eddo in ekkatak in Dr. Pearl McElfish ilo 479-713-8680 ak ilo pamcelfish@uams.edu, elañe Please call the head researcher of the study Dr. Pearl McElfish at 479-713-8680 if you
  - ✓ ewor am kajjitōk ikijien ekkatak in, have any questions about this study
  - ✓ ewōr am kajjitok ikijien maroñ ko am, have questions about your rights
  - ✓ eñjake ke ewōr jorāān emōj an walok ilo am bed ilo ekkatak in, feel you have been injured in any way by being in this study
- Komaroñ in tōbar rijerbal ro an UAMS ro rej loloodjake ekkatak in ñe kwoj jab maroñ tōbar rijerbal ro ak kwoj kōnaan tōbar juon eo ejjab jerbal ilo ekkatak in. Kūr tok UAMS review board eo ilo 501-686-5667 ilo awa in jerbal ko. You can also call the office at UAMS that supervises research if you can't reach the study team or want to speak to someone not directly involved with this study. To do so call the UAMS Institutional Review Board at 501-686-5667 during normal work hours.

Organizations

PI (researcher): Pearl McElfish, PhD

# University of Arkansas for Medical Sciences HIPAA Authorization Form

- Health Insurance Portability and Accountability Act of 1996 ej kakien eo an United States im ej komman kakien ko ikijien kojbarok melele in takto ko an armij. Health Insurance Portability and Accountability Act of 1996 is the United States legislation that provides data privacy and security provisions for safeguarding medical information.
- Naan eo "kwe" ej jerbal ñan melele kein ruo: armij eo ej bōk konaan ilo ekkatak in koba armij eo ej letok mālim in bed ilo ekkatak in. Pepa in koba pepa in mālim eo (consent form) rej aikuj koba ibben dron ilo aer lewaj melele kein. The word "you" means both the person who takes part in the research study. This form and the program consent form need to be kept together.

Jej kajitok bwe kwon bōk konaam ilo ekkatak in im emōj kōmeleleiki ilo pepa in consent form ak mālim eo. Ñan kōmmane ekkatak in, jenaj aikuj bōk melele ko rej kallikar wōn kwe. Jemaron naaj kajjitōk kōn melele kein:

- raan in lōtak
- kōrā/emmaan
- emōj ke mare
- jete armij ilo kabijuknen eo am
- jikuul
- jerbal
- injuren
- Nañinmej ko jet remaron walok jen nañinmej in tōñal
- taktō
- kwoj jen ia/lal eo am
- aitokam
- eddoim
- bororo
- kakōlkōl ko nan naninmij in tōnal
- kakōlkōl ko nan naninmij in kūriij
- blood pressure ak aibōlat
- jiban jen baamle eo
- kōjbarok am eddo
- exercise ak makūtkūt
- kain mōnā im dren ko nimōm
- wā in COVID19 ko am

Organizations

PI (researcher): Pearl McElfish, PhD

• uno ko kwōj būki

Melele kein renaj kōjerbali ñan kōlablok melele ko ad ikkijien kōmman kilaaj kōn nañinmij in tônal im wāwein kōjbarok. Jenaaj bōk wōt melele ko jej aikuji ñan ekkatak in. Melele ko renaaj walok ilo am bôk konaam ilo ekkatak in rej einwōt:

- jonan juka ak tonal eo ilo anbwinnum
- joñan aer in bōtōktōk ilo ānbwinnūm

Bwe kwon bed ilo ekkatak in, kwoj aikuj letok mãlim bwe jen bõk melele ko am, kōbooji, im je pepa ko nan kwalok tōbrak in ekkatak in.

Kōm naaj, ak kōm maroñ kwalok melele kōn ejmour eo am ibben armij ro ilo University of Arkansas for Medical Sciences (UAMS) ro im rej jibañ kōn ekkatak in, einwōt rijerbal ro an ekkatak in, UAMS Institutional Review Board eo, im obiij eo ej bōk eddoin kakien ko an ekkatak ko ilo UAMS.

Kom maroñ kwalok melele ko ikijien ejmour eo am ibben armij ro itulikin UAMS im rej loloorjake bwe en jimwe ad kōmmani ekkatak kein, einwōt obiij eo an Office for Human Research Protections im obiij ko rej bar loloorjake ak koba lok ibbeir ilo aer jerbali kakien kein an ekkatak in. Jej kōtmene bwe ro rej bōk konaer ilo kōmmani ekkatak ko remelele aurōkin kōjbarok melele ko am. Bōtaab, jet armij ro itulikin in UAMS remaroñ lilok melele ko am ñan bar jet. Elañe renaaj, kakien eo UAMS ej aikuj loore remaroñ jab jelet er im remaroñ jab kōjbarok melele ko am.

Pepa in mālim in nān bōk, kōjerbal, im lelok melele ko am enaaj jemlok kitien ilo ien eo ejemlok ekkatak in. Ilo jemlok in pepa in, komaron kelet bwe jen bar kojerbal melele ko am nān ekkatak ko iliju im jeklaj.

Elañe kwonaaj jaini pepa in, kwoj letok mālim bwe jen kōmman, aini im aji melele ko emōj kallikari ijin. Kwōjjab aikuj jaini pepa in. Bōtaap, elañe kwoj kelet in jab jaini pepa in, innem kwōjjab maron bed ilo ekkatak in. Kwōj aikuj jaini pepa im mālim in elañe kwōj kōnaan bed ilo ekkatak in.

Elañe kwōnaj jaini pepa in innem tokālik kallikar ke kwōjjab kōnaan bwe jen bōk ak aji melele ko am, kwōj aikuj je im jilkinlok juōn am leta ñan eo ej bōk eddoin ekkatak in ak Prinicipal Investigator eo:

Pearl McElfish, PhD University of Arkansas for Medical Sciences Northwest 2708 S 48<sup>th</sup> Street Springdale, AR 72762

Organizations

PI (researcher): Pearl McElfish, PhD

#### pamcelfish@uams.edu

Kwōnaaj aikuj jaini leta in, je etan taitōl eo an ekkatak in ie im ej bed itulōn tata in pepa in ālikin naan kein "Study Title", im aikuj je im kallikar ke emōj am ukōt am lōmnak im kwōj kabōjrak mālim eo am ilo pepa in "HIPAA Research Authorization" eo. Kwōnaaj aikuj bojrak jen ekkatak in elane jejjab maron bōk im aji melele ko am. Bōtaab, bwe jen dābij wōt melele im jimwe ko an ekkatak in, jemaron naj kōjerbal wōt melele ko am emōj kar būki mokta jen an Principal Investigator eo loe leta in nan kabōjrak am bed ilo ekkatak in.

We are asking you to take part in the research study described in the consent form. To do this program, we need to collect health information that identifies you. We may collect the following information:

- date of birth
- sex
- marital status
- number of persons in your home
- education
- employment
- insurance status
- diabetes-related health conditions
- ability to access health care
- race/ethnicity
- height
- weight
- pregnancy status
- tests for diabetes
- tests for cholesterol
- blood pressure
- support from your family
- managing your weight
- exercise
- COVID-19 vaccination history
- what you eat and drink
- what medications you take

This information will be used for the purpose of learning more about teaching diabetes self-management. We will only collect information that is needed for the research. Participating in this study will provide the following health information:

- blood sugar levels
- blood pressure levels

Organizations

PI (researcher): Pearl McElfish, PhD

For you to be included in this study, we need your permission to collect, create and share this information.

We will, or may, share your health information with people at the University of Arkansas for Medical Sciences (UAMS) who help with the research or things related to the research process, such as the program staff, the UAMS Institutional Review Board and the research compliance office at the University of Arkansas for Medical Sciences.

We may need to share your health information with people outside of UAMS who make sure we do the program properly, such as the Office for Human Research Protections and other institutional oversight offices. We believe that those involved with programs understand the importance of preserving the confidentiality of your health information. However, some of the people outside of UAMS may share your health information with someone else. If they do, the same laws that UAMS must obey may not apply to others to protect your health information.

This authorization to collect, use and share your health information expires at the end of the program unless you agree to allow us to use your de-identified information for future research at the bottom of this form.

If you sign this form, you are giving us permission to create, collect, use and share your health information as described in this form. You do not have to sign this form. However, if you decide not to sign this form, you cannot be in the program. You need to sign this form and the consent form if you want to be in the program.

If you sign this form but decide later that you no longer want us to collect or share your health information, you must send a letter to Principal Investigator:

Pearl McElfish, PhD University of Arkansas for Medical Sciences Northwest 2708 S 48<sup>th</sup> Street Springdale, AR 72762 pamcelfish@uams.edu

The letter needs to be signed by you, should list the "Study Title" listed on this form, and should state that you have changed your mind and that you are revoking your "HIPAA Research Authorization". You will need to leave the program if we cannot collect and share any more health information. However, in order to maintain the reliability of the research, we may still use and share your information that was collected before the Principal Investigator received your letter withdrawing the permissions granted under this authorization.

Organizations

PI (researcher): Pearl McElfish, PhD

# Ilo aō jaini pepa in, ij kallikar ke:

# By signing the document, I am saying:

- ✓ Naij melele ke aō bebe bōk konaō ilo ekkatak in. I understand that joining this study is voluntary.
- ✓ Naij errā in bed ilo ekkatak in. I agree to be in the study.
- ✓ Juon armij ear konono ibba kōn melele ko ilo pepa in im uwaaki aōlep kajjitōk ko aō.
- ✓ Someone talked with me about the information in this document and answered all my questions.

# Ijelā ke:

### I know that:

- ✓ Imaron bojrak jabdewot ien ilo ekkatak in, im ejjelok jorāān enaaj walok nan na. I can stop any and all parts of the study at any time and nothing bad will happen to me.
- ✓ Imaroñ kūr lok obiij eo ej bõk eddo in ekkatak ko (UAMS Institutional Review Board) ilo 501-686-5667 elañe ewōr jabdewōt kajjitōk ko ikijien ekkatak in ak ikijien maroñ ko aõ. I can call the office that supervises research (UAMS Institutional Review Board) at 501-686-5667 if I have any questions about the study or about my rights.
- ✓ Ijjab julok maron ko aō ilo aō jaini pepa in. I do not give up any of my rights by signing this form.
- ✓ Kelet eo ao eban kōmman oktak ilo aō nej etal wōt n̄an UAMS in taktō. My decision will not change my medical care at UAMS.

| Naij errā in bed ilo ekkatak in. |
|---|
| I agree to be part of this study. |
| ☐ YES/AET ☐ NO/JAAB |
| Ij lelok mālim bwe UAMS en kōjerbal melele ko aō ilo ekkatak nan ekkatak ko jet UAMS ej kōmmani. |
| I give permission for UAMS to link information from this study to other studies conducted by UAMS. |
| ☐ YES/AET ☐ NO/JAAB |
| Ij errā bwe melele ko aō im emoj jolok etta jeni ren wōnmaanlok wōt im kojerbali n̄an ekkatak ko an tōn̄al iliju im jōklaj. |
| I agree to my de-identified information being used for future diabetes-related research. |

| Organizations PI (researcher): Parling Model of Diabetes Sell-I Pa | | -Management Education in Faith Based |
|---|---|---|
| YES/AET NO | O/JAAB | |
| _ | | |
| Ij errā bwe ren kenaanik āa ikijien ekkatak ko jet iliju im jōklaj. I agree to being contacted for future research related to this study. | | |
| Etam (jouj im kallikare) | | Jaini etam |
| Your name (please print) | | Your signature |
| | | Ç |
| Raan eo | | |
| Date | | |
| Armej eo ej loloodjake mālim in ( kallikar etam) | | Jain eo an armej eo ej loloodjake mālim in |
| Person Obtaining Consent name (please print) | | Person Obtaining Consent signature |
| Raan eo | | |
| Date | | |